CLINICAL TRIAL: NCT04486885
Title: European Study of Cerebral Aspergillosis Treated With Isavuconazole
Acronym: ESCAI
Status: Completed | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: hj-20-ESCAI
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Aspergillosis; Invasive Aspergillosis
Keywords: cerebral aspergillosis; isavuconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study clinical context Cerebral aspergillosis (CA) is a rare location of invasive aspergillosis (IA), associated with a high morbidity and mortality. Since 2002, voriconazole is the recommended first line treatment of invasive aspergillosis. More recently, isavuconazole appeared to be not less effective than voriconazole in the treatment of filamentous IFI, with a better tolerance profile.

The investigators aim to evaluate better the efficacy and the safety of isavuconazole in the treatment of cerebral aspergillosis by a descriptive, multicentric, international retrospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Proven or probable cerebral aspergillosis according to the EORTC criteria modified by adding diabetes in the host criteria
* In child or adult
* Treated by isavuconazole at least 7 days
* Diagnosed between March 2017 and June 2020

Exclusion Criteria:

* Possible cerebral aspergillosis
* isavuconazole treatment for less than 7 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 40 adult ou pediatric patients, suffering frome cerebral aspergillosis, diagnosed between 2017 and 2020, and treated by isavuconazole at least 7 days
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Outcome of the patients : alive without CA treatment/alive under CA treatment/ deceased. | At baseline
  Number of patients alive without CA treatment/alive under CA treatment/ deceased.

SECONDARY OUTCOMES:
Monitoring of isavuconazole : dosage in the serum and in the cerebro-spinal-fluid | At baseline
  dosage of isavuconazole in the serum and in the cerebro-spinal-fluid
-Adverse events under isavuconazole and drug interactions | At baseline
  Adverse events under isavuconazole and drug interactions

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Lanternier, MD, Principal Investigator — Hôpital Necker
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France